CLINICAL TRIAL: NCT05928559
Title: The Relationship Between Body Composition and Physical Fitness in Young Male Basketball Players
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Gökhan Can TÖRPÜ, Principal Investigator, Bezmialem Vakif University
Other Study IDs: BezmialemVU-KFR-GCT-01
Record Dates: First submitted 2023-06-15; First posted 2023-07-03 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sports Physical Therapy
Keywords: Basketball; Body Composition; Aerobic Capacity; Muscle Endurance; Muscle Strenght

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Male Basketball Players: Male athletes between the ages of 10-24 who are involved in a local basketball academy and have been involved in basketball for more than a year
  Interventions: Other: OMRON BF511 Body Composition Monitor

INTERVENTIONS:
Other: OMRON BF511 Body Composition Monitor — The OMRON BF511 Body Composition Monitor is a digital scale and participants' body compositions will be evaluated with this device. The aerobic capacities of the participants will be evaluated with the Multi-Stage 20 m Shuttle Run Test and the maximum oxygen consumption levels will be calculated with the help of the formula with the data obtained from this test. The trunk extensor muscle endurance of the participants will be evaluated with the Biering-Sorensen Test and the trunk flexor endurance will be evaluated with the Kraus-Weber Test. Participants' M. Quadriceps, M. Hamstring, M. Biceps Brachii and M. Triceps Brachii muscle strengths will be evaluated with MicroFET® 2 hand dynamometer.
  Other Names: Multi-Stage 20 m Shuttle Run Test; Biering-Sorensen Test and Kraus-Weber Test; MicroFET® 2 hand dynamometer

SUMMARY:
In this study, it is aimed to investigate the relationship between body composition, aerobic capacity, trunk muscle endurance and muscle strength in young male basketball players.

The study will take place at a local basketball academy. Young male athletes between the ages of 10-24 and enrolled in a basketball academy will be included in the study. Participants who have been involved in basketball for less than a year, and those who have injuries that prevent participation in the study will be excluded.

DETAILED DESCRIPTION:
Individual development differences in young people can have an impact on physical fitness components such as aerobic capacity, trunk muscle endurance and muscle strength required for basketball. At the same time, differences in these components can have effects on each other.

There is a complex relationship between anthropometric changes during growth and physical fitness because many differences can occur during the physiological development of players. In this context, differences in growth rate and development in young basketball players are complex factors that affect game performance and player success. Characteristics such as body height, body weight, skeletal muscle ratio and body fat are among the basic anthropometric components of a basketball player, and these components are considered to be important indicators of a player's game performance.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Being between the ages of 10-24

Exclusion Criteria:

* Athlete's own or family refusal to participate in the study
* Interested in basketball for less than a year
* Having an injury that would prevent participation in the study

Ages: 10 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Young male basketball players enrolled in a local basketball academy
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Body Weight | One Month
  Participants' body weights will be evaluated with the OMRON BF511 Body Composition Monitor and recorded in kilograms (kg).
Body Height | One Month
  The body lengths of the participants will be evaluated with a tape measure and recorded in meters (m).
Body Mass Index | One Month
  The body mass index of the participants will be calculated and recorded with the formula kg/m^2.
Body Fat | One Month
  Participants' body fat will be evaluated with the OMRON BF511 Body Composition Monitor and recorded in percent (%).
Skeletal Muscle Mass | One Month
  Participants' skeletal muscle mass will be evaluated with the OMRON BF511 Body Composition Monitor and recorded in percent (%).
Visceral Fat | One Month
  Participants' visceral fat will be evaluated with the OMRON BF511 Body Composition Monitor and recorded in levels.
Resting Metabolic Rate | One Month
  Participants' visceral fat will be evaluated with the OMRON BF511 Body Composition Monitor and recorded in kilocalories (kcal).
Aerobic Capacity | One Month
  Maximum oxygen consumption (VO2max)
Trunk Muscle Endurance | One Month
  Trunk extensor muscle endurance will be evaluated with Biering-Sorensen Test and trunk flexor muscle endurance will be evaluated with Kraus-Weber Test. The maximum time the participants can continue the test will be recorded in seconds.
Muscle Strength | One Month
  M. Quadriceps, M. Hamstring, M. Biceps Brachii and M. Triceps Brachii muscles will be evaluated in Newtons (N) with MicroFET® 2 hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan C Törpü, BPT, Principal Investigator — Bezmialem Vakif University; Semiramis Özyılmaz, PhD, Study Director — Bezmialem Vakif University; Selva Otsay, BPT, Study Chair — Bezmialem Vakif University
Locations (1):
- Eyüp Basket Akademi, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rinaldo N, Toselli S, Gualdi-Russo E, Zedda N, Zaccagni L. Effects of Anthropometric Growth and Basketball Experience on Physical Performance in Pre-Adolescent Male Players. Int J Environ Res Public Health. 2020 Mar 25;17(7):2196. doi: 10.3390/ijerph17072196. PMID 32218293
- [Result] Toselli S, Campa F, Maietta Latessa P, Greco G, Loi A, Grigoletto A, Zaccagni L. Differences in Maturity and Anthropometric and Morphological Characteristics among Young Male Basketball and Soccer Players and Non-Players. Int J Environ Res Public Health. 2021 Apr 8;18(8):3902. doi: 10.3390/ijerph18083902. PMID 33917743